CLINICAL TRIAL: NCT04583813
Title: Efficacy of Empagliflozin in Patients With Heart Failure and Atrial Fibrillation
Brief Title: Empagliflozin and Atrial Fibrillation Treatment
Acronym: EMPA-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Massimo Grimaldi, Head of Arrhythmology and Electrophysiology Unit, Miulli General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MGH_001
Record Dates: First submitted 2020-07-20; First posted 2020-10-12 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation; Heart Failure; Obesity; Diabetes Mellitus
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Obesity; Diabetes Mellitus | interventions — empagliflozin; Tablets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): Empagliflozin 10 mg oral tablet, once daily, for 24 months
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Empagliflozin matching placebo oral tablet, once daily for 24 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 10 mg oral tablet, once daily, for 24 months
  Other Names: Empagliflozin 10 mg oral tablet
  Arms: Empagliflozin
Other: Placebo — Empagliflozin matching placebo, once daily, for 24 months
  Other Names: Placebo oral tablet
  Arms: Placebo

SUMMARY:
The primary purpose of this trial is to evaluate the impact of empagliflozin, as compared with placebo, in patients with diabetes mellitus or overweight, heart failure and atrial fibrillation.

DETAILED DESCRIPTION:
A 24-month randomized, single-blind, placebo-controlled trial to investigate the efficacy of empagliflozin to reduce atrial fibrillation burden in patients with diabetes mellitus or overweight, heart failure and atrial fibrillation in which a rhythm control strategy is indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Diabetes mellitus or Body Mass Index over 25 Kg/m2
3. Heart failure
4. New York Heart Association (NYHA) Functional Classification: II or III
5. Documented atrial fibrillation
6. Understands the nature of the study, treatment procedure and provides written informed consent
7. Willing to comply with specified pre-, post- and follow-up testing, evaluations and requirements
8. Expected to remain available for at least 24 months after enrollment

Exclusion Criteria:

1. Permanent atrial fibrillation
2. Current use or prior use of a sodium-glucose co-transporter (SGLT) 2 inhibitor or combined inhibitor of SGLT-1 and SGLT-2 (all the other antidiabetic drugs are permitted performing an accurate glycemic control)
3. Known allergy or hypersensitivity to any SGLT-2 inhibitors
4. History of ketoacidosis
5. Need or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
6. New York Heart Association (NYHA) Functional Classification: I or IV
7. Unstable angina
8. Presence of any disease that is likely to shorten life expectancy to < 1 year
9. Any cardiac surgery within three months prior to enrolment
10. Awaiting cardiac transplantation or other cardiac surgery within the next year
11. Myocardial infarction within 60 days prior to enrolment
12. Contraindications to oral anticoagulation
13. Active systemic infection or sepsis
14. Left atrial thrombus (e.g., transesophageal echocardiography, computed tomography and intracardiac echocardiography)
15. History of a documented thromboembolic event such as stroke or transient ischemic neurological attack in the three months prior to enrollment
16. Currently enrolled in another trial that has not completed the required follow-up period and would conflict with this study
17. Chronic liver diseases
18. Chronic kidney disease (creatinine clearance < 45 ml/min)
19. Pregnant or breast-feeding mothers
20. Any other clinical condition that might jeopardize patient safety during participation in this trial or prevent the subject from adhering to the trial protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Maintenance of sinus rhythm after the blanking period | From 90 days after baseline to 24-months
  To compare the proportion of patients with sinus rhythm from 90 days after baseline to end of study period

SECONDARY OUTCOMES:
Composite of major adverse cardiovascular events | Baseline through 24-months
  To compare the incidence at the end of study period of major adverse cardiovascular events (death, non-fatal myocardial infarction, acute cerebrovascular events)
Hospitalizations for cardiovascular events | Baseline through 24-months
  To compare the incidence at the end of study period of hospitalizations for cardiovascular events
Safety endpoint: Incidence of adverse events | Baseline through 24-months
  To estimate the incidence of adverse events

OTHER OUTCOMES:
Economic burden of hospitalizations for cardiovascular events | Baseline through 24-months
  To compare economic burden of hospitalizations for cardiovascular events estimated as the hospital reimbursement from National Health Service for cardiovascular admissions during study period
Changes in measure of the adverse effects of heart failure on patient's life | Baseline, 1, 3, 6, 12 and 24 month
  To compare changes in adverse effects of heart failure on patient's life evaluated by using the Minnesota Living with Heart Failure Questionnaire. The total score range is 0 to 105, with higher scores indicating more significant impairment in health-related quality of life. A total score decrease indicates the amelioration of the quality of life.
Changes in patient's perception of health status | Baseline, 1, 3, 6, 12 and 24 month
  To compare changes in perception of health status evaluated by using the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12). The total score range is 0 to 100, with higher scores indicating a better condition. A total score increase indicates amelioration of quality of life.
Changes in patient's functional capacity | Baseline, 1, 3, 6, 12 and 24 month
  To compare changes in functional capacity evaluated by using the Six Minutes Walk Test. The distance covered over a time of 6 minutes measures functional capacity. An increase in the distance walked indicates improvement in the patient's condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Miulli General Hospital, Acquaviva delle Fonti, Bari, Italy